CLINICAL TRIAL: NCT01414101
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose, Phase 2 Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ISIS 329993 in Subjects With Rheumatoid Arthritis
Brief Title: Safety, Tolerability, and Pharmacodynamic Study of ISIS CRP Rx in Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISIS 329993-CS3
Record Dates: First submitted 2011-07-21; First posted 2011-08-11 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ISIS 329993

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): Dose 1 ISIS CRP Rx versus Placebo
  Interventions: Drug: ISIS CRP Rx or Placebo
- Group B (Experimental): Dose 2 ISIS CRP Rx versus Placebo
  Interventions: Drug: ISIS CRP Rx or Placebo
- Group C (Experimental): Dose 3 ISIS CRP Rx versus Placebo
  Interventions: Drug: ISIS CRP Rx or Placebo

INTERVENTIONS:
Drug: ISIS CRP Rx or Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of ISIS CRP Rx and its effects on CRP and other pharmacodynamic measures, versus placebo, in subjects with active rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female; age 18 to 75 years
* Active RA for at least 6 months
* Active disease defined by having equal to or greater than 6 swollen joints and 6 tender joints, based on a 28 joint count
* On stable doses and regimen of allowed RA medications
* Currently receiving at least 10 mg of methotrexate a week. Patients unable to tolerate doses greater than 10 mg may also be eligible for enrollment.

Exclusion Criteria:

* Diagnosis of Felty's syndrome, psoriatic arthritis, gout, or auto-immune rheumatic disease
* Any surgical procedure within 30 days of Screening or likely to need joint or tendon surgery or other surgical procedure during the study
* Intra-articular or intra-muscular corticosteroids within 60 days prior to dosing
* Previous treatment with any biologic response modifying agent for RA within 90 days or 5 half-lives, whichever is greater, prior to screening
* Previous treatment with rituximab at any time
* Use of corticosteroid therapy equivalent to an average daily dose of >10 mg of prednisone
* Any Screening laboratory values that are out of allowed reference ranges
* Inability to comply with protocol or study procedures
* Any other significant illness or condition that may adversely affect the subjects participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Safety | 155 Days
  Adverse events, laboratory tests, and vital signs

SECONDARY OUTCOMES:
hsCRP | 155 Days
  The effects of treatment with ISIS CRP Rx or Placebo on hsCRP

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (3):
  - Isis Investigational site, Kamloops, British Columbia
  - Isis Investigational Site, Toronto, Ontario
  - Isis Investigational Site, Montreal, Quebec
- Russia (2):
  - Isis Investigational Site, Moscow
  - Isis Investigational Site, Saint Petersburg

REFERENCES:
- [Derived] Warren MS, Hughes SG, Singleton W, Yamashita M, Genovese MC. Results of a proof of concept, double-blind, randomized trial of a second generation antisense oligonucleotide targeting high-sensitivity C-reactive protein (hs-CRP) in rheumatoid arthritis. Arthritis Res Ther. 2015 Mar 19;17(1):80. doi: 10.1186/s13075-015-0578-5. PMID 25885521